CLINICAL TRIAL: NCT05168189
Title: Ivabradine and Its Role in the Development of Atrial Fibrillation in Patients With Chronic Coronary Syndrome
Brief Title: the Role of Ivabradine in Causing AF in Patients With Chronic Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ragab Kamel, Resident doctor, Assiut University
Other Study IDs: Ivabradine-induced AF in CCS
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: AF - Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ivabradine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | US Export: No

GROUPS / COHORTS (2):
- Ivabradine Group: patients with chronic coronary syndrome using Ivabradine for heart rate control or as anti-anginal treatment.
  Interventions: Drug: Ivabradine; Diagnostic Test: transthoracic echo; Device: 24 hours holter
- Non-Ivabradine Group: patients with chronic coronary syndrome NOT using Ivabradine for heart rate control or as anti-anginal treatment.
  Interventions: Diagnostic Test: transthoracic echo; Device: 24 hours holter

INTERVENTIONS:
Drug: Ivabradine — follow up chronic coronary syndrome patients receiving Ivabradine for ( 6 months ) if the participants develop atrial fibrillation using 24 hours holter .
  Other Names: Procoralan , Corlanor,
  Groups: Ivabradine Group
Diagnostic Test: transthoracic echo — performing baseline transthoracic echo for all patients to exclude any chamber dilatation
  Other Names: TTE
Device: 24 hours holter — perform 24 hours Holter monitoring for all patients at the start of the study and follow up after 6 months

SUMMARY:
This study is aiming to detect the possibility of Ivabradine's role in the development of atrial fibrillation in chronic coronary syndrome patients with No structural heart disease.

DETAILED DESCRIPTION:
Ivabradine is a heart rate-lowering agent best characterized by its negative chronotropic effect on the sinoatrial node. Its unique mechanism selectively blocks the pacemaker funny channels, which are responsible for spontaneous depolarization in the sinoatrial node that regulates heart rate during sinus rhythm. It has been well established that controlling the heart rate is the main target when treating coronary artery disease and heart failure and is associated with a beneficial effect on mortality and morbidity.

According to the European Society of Cardiology guidelines for Chronic coronary syndrome, ivabradine should be considered as an anti-anginal agent in patients with sinus rhythm and heart rate of ≥70 BPM in combination with beta-blockers or when beta-blockers are not tolerated.

The If current, which is affected by ivabradine, was found to be present in the pulmonary vein myocardial sleeves, the well-recognized triggers for AF.

This may explain the risk of AF in patients receiving this drug. However, AF is commonly associated with HF and ischemic heart disease, the current two clinical indications for the use of ivabradine, hence AF in this patient population may be an association rather than a drug-induced effect.

Previously, ivabradine's heart rate reduction was thought to be exclusively due to inhibition of If channels in the sinoatrial node. However, emerging data have shown channels that maintain the If current in the free wall of both atria. These findings support the idea that the If current plays a role in the pathophysiological procedure that initiates and maintains AF.

ELIGIBILITY:
Inclusion Criteria:

* age range from 18 to 70 years.
* diagnosed with Chronic Coronary syndrome according to European association guidelines of 2019.
* Normal structural heart disease (as evident by 2D transthoracic echocardiography).
* in sinus rhythm.

Exclusion Criteria:

* Patient with heart rate below 70 bpm at the start of treatment.
* Smokers.
* hyperthyroidism.
* Hypertensive patients
* Patient with bradycardia arrhythmia (sinus Bradycardia, advanced degree of heart block).
* history of Atrial fibrillation.
* history of Myocardial infarction, Previous PCI, or CABG.
* Patient with Valvular heart disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic coronary syndrome attending an outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
detect the incidence of Ivabradine-induced AF in patients with chronic coronary syndrome | 6 months after the start of Ivabradine treatment
  detect the role of Ivabradine's in the development of atrial fibrillation in chronic coronary syndrome patients with No structural heart disease.

CONTACTS AND LOCATIONS:
Overall Officials: Salwa R. Demitry, PhD, Study Director — Professor at cardiovascular medicine department , assiut university

REFERENCES:
- [Background] Koruth JS, Lala A, Pinney S, Reddy VY, Dukkipati SR. The Clinical Use of Ivabradine. J Am Coll Cardiol. 2017 Oct 3;70(14):1777-1784. doi: 10.1016/j.jacc.2017.08.038. PMID 28958335
- [Background] DiFrancesco D. Funny channels in the control of cardiac rhythm and mode of action of selective blockers. Pharmacol Res. 2006 May;53(5):399-406. doi: 10.1016/j.phrs.2006.03.006. Epub 2006 Mar 27. PMID 16638640
- [Background] Dyer AR, Persky V, Stamler J, Paul O, Shekelle RB, Berkson DM, Lepper M, Schoenberger JA, Lindberg HA. Heart rate as a prognostic factor for coronary heart disease and mortality: findings in three Chicago epidemiologic studies. Am J Epidemiol. 1980 Dec;112(6):736-49. doi: 10.1093/oxfordjournals.aje.a113046. PMID 7457467
- [Background] Kannel WB, Kannel C, Paffenbarger RS Jr, Cupples LA. Heart rate and cardiovascular mortality: the Framingham Study. Am Heart J. 1987 Jun;113(6):1489-94. doi: 10.1016/0002-8703(87)90666-1. PMID 3591616
- [Background] Hoppe UC, Beuckelmann DJ. Characterization of the hyperpolarization-activated inward current in isolated human atrial myocytes. Cardiovasc Res. 1998 Jun;38(3):788-801. doi: 10.1016/s0008-6363(98)00047-9. PMID 9747448
- [Background] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Background] Suenari K, Cheng CC, Chen YC, Lin YK, Nakano Y, Kihara Y, Chen SA, Chen YJ. Effects of ivabradine on the pulmonary vein electrical activity and modulation of pacemaker currents and calcium homeostasis. J Cardiovasc Electrophysiol. 2012 Feb;23(2):200-6. doi: 10.1111/j.1540-8167.2011.02173.x. Epub 2011 Sep 13. PMID 21914029
- [Background] Abdelnabi M, Ahmed A, Almaghraby A, Saleh Y, Badran H. Ivabradine and AF: Coincidence, Correlation or a New Treatment? Arrhythm Electrophysiol Rev. 2020 Feb 12;8(4):300-303. doi: 10.15420/aer.2019.30.2. PMID 32685161
- [Background] Salaria V, Mehta NJ, Abdul-Aziz S, Mohiuddin SM, Khan IA. Role of postoperative use of adrenergic drugs in occurrence of atrial fibrillation after cardiac surgery. Clin Cardiol. 2005 Mar;28(3):131-5. doi: 10.1002/clc.4960280306. PMID 15813619